CLINICAL TRIAL: NCT01525966
Title: Phase II Trial of Neoadjuvant Chemotherapy With Carboplatin and NAB-Paclitaxel in Patients With Locally Advanced and Inflammatory Triple Negative Breast Cancer
Brief Title: Carboplatin and Paclitaxel Albumin-Stabilized Nanoparticle Formulation Before Surgery in Treating Patients With Locally Advanced or Inflammatory Triple Negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11174; NCI-2012-00025 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-01-27; First posted 2012-02-03 (Estimated); Results first posted 2023-03-10 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Inflammatory Breast Cancer; Stage IIA Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Triple-negative Breast Cancer; Stage IIB Breast Cancer; Estrogen Receptor Negative; Progesterone Receptor Negative; HER2/Neu Negative
MeSH Terms: conditions — Inflammatory Breast Neoplasms; Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Carboplatin; Taxes; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (carboplatin and nab-paclitaxel) (Experimental): Patients receive carboplatin IV over 30 minutes on day 1 and paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes once weekly. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: carboplatin; Drug: paclitaxel albumin-stabilized nanoparticle formulation; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Drug: paclitaxel albumin-stabilized nanoparticle formulation — Given IV
  Other Names: ABI-007; nab paclitaxel; nab-paclitaxel; nanoparticle albumin-bound paclitaxel
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well carboplatin and nab-paclitaxel before surgery work in treating patients with triple negative breast cancer that is inflammatory or has spread from where it started to nearby tissue or lymph nodes. Drugs used in chemotherapy, such as carboplatin and nab-paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test the hypothesis that carboplatin + nab-paclitaxel (paclitaxel albumin-stabilized nanoparticle formulation) therapy will demonstrate a promising neoadjuvant pathologic complete response (pCR) rate for eligible patients.

II. To test the hypothesis that carboplatin + nab-paclitaxel therapy will demonstrate a promising Symmans 0-1 pathological response rate for eligible patients.

SECONDARY OBJECTIVES:

I To evaluate the overall survival and event-free survival of eligible patients treated with carboplatin + nab-paclitaxel neoadjuvant chemotherapy.

II. To evaluate the toxicities and tolerance of carboplatin + nab-paclitaxel therapy in this patient population.

III. To evaluate the role of laboratory correlates in response, toxicity and survival endpoints.

IV. To procure tissue and perform analysis of gene and protein expression profiles of pre-treatment primary tumor (estimated success rate: 80%) and residual tumors (25%) and lymph nodes including the study of tumor niche (50%), studying sequential assessment of cellular characteristics and gene and protein expression profiles.

V. To identify specific mutations in tumor deoxyribonucleic acid (DNA) in comparison to adjacent tissue and germ line DNA procured prior to, during, and subsequent to neoadjuvant chemotherapy, and to detect/measure, as feasible, the presence of such mutations in fragmented circulating DNA from plasma, and to correlate these mutations with the presence/characteristics of circulating tumor cells in order to identify prognostic and predictive indicators of persisting/relapsed disease and targets for therapy.

VI. To assess ribonucleic acid (RNA) (using Mammaprint/Blueprint and 44,000 Agilent platform gene array), (micro) miRNA and exosome and protein profiles in tumor, adjacent tissue and plasma prior to, during, and at completion of neoadjuvant chemotherapy in order to establish prognostic and predictive indicators of outcome, markers of persistent/relapsed disease, and targets for therapy.

VII. To analyze tumor DNA and genomic DNA from plasma by microarray and reverse transcriptase (RT)-polymerase chain reaction (PCR) analysis to assess copy numbers/single nucleotide polymorphisms (SNP)/genomic polymorphisms in genes for the purposes of establishing prognostic and predictive indicators of outcomes; markers of persistence/relapse disease, drug resistance, and drug metabolism; and targets of therapy.

VIII. To assess the prognostic and predictive value of conventional pathological features (stage, estrogen and progesterone receptor and human epidermal growth factor receptor [HER-2] status, presence of lymphovascular invasion, high grade tumor status) in comparison to such values derived from the molecular approaches.

IX. To procure tumor from the primary and definitive surgical specimen for the purpose of establishing breast cancer stem cell lines.

X. To procure blood samples for the purpose of identifying and characterizing circulating tumor cells.

OUTLINE: Patients receive carboplatin intravenously (IV) over 30 minutes on day 1 and paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes once weekly. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 4 years and then every 6 months for 1 year and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be diagnosed with locally advanced (T2 and higher with or without lymph node involvement), and/or inflammatory triple negative breast cancer
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* Tumor negative for expression of hormone receptors (< 10%) and not over-expressing HER2 by immunohistochemistry (IHC) (0-1), or in case of IHC of 2, negative by fluorescence in situ hybridization (FISH) or by alternative gene testing
* Bilirubin =< 1.5 mg/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2 x upper limit of normal
* Alkaline phosphatase =< 2 x upper limit of normal
* Platelets >= 100,000 cells/mm^3
* Hemoglobin > 9.0 g/dL
* Absolute neutrophil count (ANC) >= 1,500 cells/mm^3
* Creatinine =< 1.5 mg/dL is recommended; however, institutional norms are acceptable
* Left ventricular ejection fraction > 50%
* Women of childbearing potential and sexually active males must use an effective contraception method during treatment and for three months after completing treatment
* Negative serum or urine beta-human chorionic gonadotropin (hCG) pregnancy test screening for patients of childbearing potential
* All subjects must have the ability to understand and the willingness to sign a written informed consent
* No prior therapies are allowed for the treatment of the newly diagnosed breast cancer; patients with a prior diagnosis of malignancy treated >= 5 years ago are eligible, provided that they have not received prior taxanes or carboplatin as part of their prior treatment regimen, and that they meet all eligibility criteria

Exclusion Criteria:

* Known active hepatitis B or C
* Known active human immunodeficiency virus (HIV)
* Prior breast cancer or other invasive malignancy treated within 5 years
* Pregnancy
* Neuropathy > grade 1
* Any other intercurrent medical/psychological problem deemed exclusionary by the treating physician or investigators/primary investigator (PI)
* Subjects will be excluded who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2012-02-15 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2025-12-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Mortimer, MD, PhD, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - City of Hope- South Pasadena Cancer Center, South Pasadena, California

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants for this study will be recruited from among patients undergoing treatment at City of Hope Cancer Center for stage II/III -- including inflammatory-- breast adenocarcinoma. Patients will be recruited through encounters by the Breast Oncologists in the Department of Medical Oncology and/or Breast Surgical Oncologists of the Department of General Oncological Surgery.
Period: Overall Study
Arm/Group | Treatment (Carboplatin and Nab-paclitaxel)
Started | 67
Completed | 67
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Eligibility criteria included: Locally advanced (T2 and higher with or without lymph node involvement), and/or inflammatory breast cancer; triple negative biology only. Tumor negative for expression of hormone receptors (IHC < 10%) and not overexpressing HER2 by IHC (O-1), or, in case of IHC of 2, negative by FISH or by alternative gene testing. Greater than 18 years of age, female. Adequate organ function as specified in the protocol.
Arm/Group | Treatment (Carboplatin and Nab-paclitaxel)
Number analyzed (Participants) | 67
Age, Continuous [Median (Full Range); unit: years] | 52 [28 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 35
  Hispanic | 24
  Asian | 4
  African American | 1
  Other | 3
Region of Enrollment [Number; unit: participants]
  United States | 67

OUTCOME MEASURES:

1. Primary Outcome: pCR Rate After Treatment.
Description: pCR is RCB 0 by Symmans criteria. The goal of the study is a detection of an increase in rate of pathological complete remission (pCR) from 20% (historical) to 38%
Time Frame: At completion of definitive surgery, up to six months from initial treatment
Population: Sixty-seven patients met the eligibility criteria for inclusion in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Carboplatin and Nab-paclitaxel)
Number analyzed (Participants) | 67
Participants
  pCR | 32
  not reached pCR | 35

2. Primary Outcome: Residual Cancer Burden (RCB) by Symmans Criteria.
Description: Categorization of the outcome of the treatment at completion of definitive surgery by Symmans criteria. "The index score is derived from the largest area and cellularity of residual invasive primary cancer and the number of involved lymph nodes and size of largest metastasis. pCR (stage yp-T0/is, ypN0) has RCB = 0; and RCB class is minimal (RCB-I), moderate (RCB-II), or extensive (RCB-III), on the basis of predefined cut points of 1.36 and 3.28 index scores.) Symmans WF, Wei C, Gould R, et al. J Clin Oncol 35:1049-1060, 2017. Symmans WF, Peintinger F, Hatzis C et al. J Clin Oncol 25:4414-4422, 2007. Order of scale is RCB0 is best, then I, II, III, worse; progressive is the worst.
Time Frame: At completion of definitive surgery, up to six months post-commencement of study chemotherapy.
Population: Sixty-seven patients met the eligibility criteria for inclusion in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Carboplatin and Nab-paclitaxel)
Number analyzed (Participants) | 67
Participants
  achieved pCR (RCB 0); no residual disease | 32
  had RCB I; minimal residual disease | 10
  had RCB II; moderate residual disease | 19
  had RCB III; extensive residual disease | 5
  Progressed | 1

3. Secondary Outcome: Adjuvant Radiation
Description: After adjuvant chemotherapy and before surgery, some patients were given adjuvant radiation.
Time Frame: Up to 6 months
Population: Sixty-seven patients met the eligibility criteria for inclusion in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Carboplatin and Nab-paclitaxel)
Number analyzed (Participants) | 67
Participants
  Radiation before surgery | 37
  No radiation was given before surgery | 29
  No radiation and no surgery | 1

4. Secondary Outcome: Scope of Surgery
Description: After having received adjuvant chemotherapy, and possibly radiation, patients underwent surgery.
Time Frame: Up to 6 months.
Population: Patients eligible for this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Carboplatin and Nab-paclitaxel)
Number analyzed (Participants) | 67
Participants
  Lumpectomy | 19
  Mastectomy | 47
  No surgery performed due to distant metastasis | 1

5. Secondary Outcome: Overall Survival
Description: Estimated by the Kaplan-Meier method. Three-year point estimate and 95% confidence interval based on the Greenwood variance, with log-log transformation, will be provided. The corresponding median survival times (with 90% confidence limits) will be determined. Patients' survival times will be measured from the initial date of treatment to the recorded date of death, or most recent follow-up at the end-of-study date.
Time Frame: Up to three years post-commencement of chemotherapy.
Population: Sixty-seven patients met the eligibility criteria for inclusion in this study.
Measure: Number (95% Confidence Interval); unit: percentage of surviving patients: 3-yr
Arm/Group | Treatment (Carboplatin and Nab-paclitaxel)
Number analyzed (Participants) | 67
percentage of surviving patients: 3-yr | 90.2 [77.8 to 95.8]

6. Secondary Outcome: Progression-free Survival
Description: Estimated by the Kaplan-Meier method. Three-year point estimate and 95% confidence interval based on the Greenwood variance, with log-log transformation, will be provided. Patients' survival times will be measured from the initial date of treatment to the recorded date of progression or death. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to three years.
Population: Sixty-seven patients met the eligibility criteria for inclusion in this study.
Measure: Number (95% Confidence Interval); unit: percentage of pts
Arm/Group | Treatment (Carboplatin and Nab-paclitaxel)
Number analyzed (Participants) | 67
percentage of pts | 87.3 [58.5 to 90.2]

ADVERSE EVENTS:
Time Frame: Serious and Other Adverse Events monitored through completion of treatment, up to 6 years, 7 months. All-Cause Mortality monitored up to 8 years.
Description: All patients eligible for this study were graded for toxicities.
Arm/Group | Treatment (Carboplatin and Nab-paclitaxel)
All-Cause Mortality (participants affected / at risk) | 5/67
Serious Adverse Events (participants affected / at risk) | 5/67
Other Adverse Events (participants affected / at risk) | 67/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Carboplatin and Nab-paclitaxel) (N=67)
10016288-Febrile neutropenia (Blood and lymphatic system disorders) | 1
10016558-Fever (General disorders) | 1
10046571-Urinary tract infection (Infections and infestations) | 1
10012174-Dehydration (Metabolism and nutrition disorders) | 2
10042613-Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Carboplatin and Nab-paclitaxel) (N=67)
10002272-Anemia (Blood and lymphatic system disorders) | 63
10016288-Febrile neutropenia (Blood and lymphatic system disorders) | 1
10007541-Cardiac disorders - Other, specify (Cardiac disorders) | 1
10019279-Heart failure (Cardiac disorders) | 1
10033557-Palpitations (Cardiac disorders) | 3
10040741-Sinus bradycardia (Cardiac disorders) | 2
10040752-Sinus tachycardia (Cardiac disorders) | 21
10061589-Aortic valve disease (Cardiac disorders) | 1
10014020-Ear pain (Ear and labyrinth disorders) | 1
10047340-Vertigo (Ear and labyrinth disorders) | 1
10065838-Middle ear inflammation (Ear and labyrinth disorders) | 1
10020705-Hyperparathyroidism (Endocrine disorders) | 1
10020850-Hyperthyroidism (Endocrine disorders) | 1
10005886-Blurred vision (Eye disorders) | 3
10010741-Conjunctivitis (Eye disorders) | 2
10013774-Dry eye (Eye disorders) | 1
10015919-Eye disorders - Other, specify (Eye disorders) | 1
10015958-Eye pain (Eye disorders) | 1
10016757-Flashing lights (Eye disorders) | 1
10016778-Floaters (Eye disorders) | 1
10047848-Watering eyes (Eye disorders) | 3
10000060-Abdominal distension (Gastrointestinal disorders) | 1
10000081-Abdominal pain (Gastrointestinal disorders) | 7
10005265-Bloating (Gastrointestinal disorders) | 1
10010774-Constipation (Gastrointestinal disorders) | 24
10012727-Diarrhea (Gastrointestinal disorders) | 16
10013781-Dry mouth (Gastrointestinal disorders) | 2
10013946-Dyspepsia (Gastrointestinal disorders) | 2
10013950-Dysphagia (Gastrointestinal disorders) | 1
10016766-Flatulence (Gastrointestinal disorders) | 2
10017947-Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2
10018286-Gingival pain (Gastrointestinal disorders) | 2
10028130-Mucositis oral (Gastrointestinal disorders) | 4
10028813-Nausea (Gastrointestinal disorders) | 40
10030980-Oral hemorrhage (Gastrointestinal disorders) | 1
10031009-Oral pain (Gastrointestinal disorders) | 4
10044055-Toothache (Gastrointestinal disorders) | 1
10047700-Vomiting (Gastrointestinal disorders) | 16
10066874-Gastroesophageal reflux disease (Gastrointestinal disorders) | 4
10008531-Chills (General disorders) | 5
10016256-Fatigue (General disorders) | 64
10016558-Fever (General disorders) | 9
10017577-Gait disturbance (General disorders) | 1
10022095-Injection site reaction (General disorders) | 1
10033371-Pain (General disorders) | 12
10050068-Edema limbs (General disorders) | 3
10062466-Localized edema (General disorders) | 4
10062501-Non-cardiac chest pain (General disorders) | 4
10001718-Allergic reaction (Immune system disorders) | 1
10002218-Anaphylaxis (Immune system disorders) | 1
10007810-Catheter related infection (Infections and infestations) | 1
10021881-Infections and infestations - Other, specify (Infections and infestations) | 2
10040872-Skin infection (Infections and infestations) | 1
10046300-Upper respiratory infection (Infections and infestations) | 7
10046571-Urinary tract infection (Infections and infestations) | 2
10055078-Bronchial infection (Infections and infestations) | 1
10061304-Nail infection (Infections and infestations) | 1
10062255-Soft tissue infection (Infections and infestations) | 1
10065772-Vulval infection (Infections and infestations) | 1
10069138-Papulopustular rash (Infections and infestations) | 1
10006504-Bruising (Injury, poisoning and procedural complications) | 3
10016173-Fall (Injury, poisoning and procedural complications) | 2
10048031-Wound dehiscence (Injury, poisoning and procedural complications) | 1
10053692-Wound complication (Injury, poisoning and procedural complications) | 1
10061103-Dermatitis radiation (Injury, poisoning and procedural complications) | 1
10001551-Alanine aminotransferase increased (Investigations) | 31
10001675-Alkaline phosphatase increased (Investigations) | 17
10003481-Aspartate aminotransferase increased (Investigations) | 24
10005364-Blood bilirubin increased (Investigations) | 4
10007839-CD4 lymphocytes decreased (Investigations) | 1
10011368-Creatinine increased (Investigations) | 7
10025256-Lymphocyte count decreased (Investigations) | 16
10029366-Neutrophil count decreased (Investigations) | 58
10035528-Platelet count decreased (Investigations) | 41
10047896-Weight gain (Investigations) | 3
10047900-Weight loss (Investigations) | 12
10049182-White blood cell decreased (Investigations) | 55
10050528-Ejection fraction decreased (Investigations) | 1
10002646-Anorexia (Metabolism and nutrition disorders) | 10
10012174-Dehydration (Metabolism and nutrition disorders) | 1
10020587-Hypercalcemia (Metabolism and nutrition disorders) | 3
10020639-Hyperglycemia (Metabolism and nutrition disorders) | 6
10020647-Hyperkalemia (Metabolism and nutrition disorders) | 2
10020670-Hypermagnesemia (Metabolism and nutrition disorders) | 1
10020680-Hypernatremia (Metabolism and nutrition disorders) | 8
10020870-Hypertriglyceridemia (Metabolism and nutrition disorders) | 5
10020943-Hypoalbuminemia (Metabolism and nutrition disorders) | 5
10020949-Hypocalcemia (Metabolism and nutrition disorders) | 10
10021005-Hypoglycemia (Metabolism and nutrition disorders) | 10
10021018-Hypokalemia (Metabolism and nutrition disorders) | 16
10021028-Hypomagnesemia (Metabolism and nutrition disorders) | 1
10021038-Hyponatremia (Metabolism and nutrition disorders) | 13
10021059-Hypophosphatemia (Metabolism and nutrition disorders) | 7
10029883-Obesity (Metabolism and nutrition disorders) | 1
10003239-Arthralgia (Musculoskeletal and connective tissue disorders) | 1
10003988-Back pain (Musculoskeletal and connective tissue disorders) | 8
10006002-Bone pain (Musculoskeletal and connective tissue disorders) | 12
10008496-Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
10016750-Flank pain (Musculoskeletal and connective tissue disorders) | 2
10028411-Myalgia (Musculoskeletal and connective tissue disorders) | 6
10028836-Neck pain (Musculoskeletal and connective tissue disorders) | 2
10031282-Osteoporosis (Musculoskeletal and connective tissue disorders) | 4
10033425-Pain in extremity (Musculoskeletal and connective tissue disorders) | 10
10062572-Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 7
10065776-Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2
10029104-Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
10045158-Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
10013573-Dizziness (Nervous system disorders) | 15
10013911-Dysgeusia (Nervous system disorders) | 5
10019211-Headache (Nervous system disorders) | 21
10027175-Memory impairment (Nervous system disorders) | 3
10029205-Nervous system disorders - Other, specify (Nervous system disorders) | 1
10029223-Neuralgia (Nervous system disorders) | 1
10033987-Paresthesia (Nervous system disorders) | 1
10034620-Peripheral sensory neuropathy (Nervous system disorders) | 53
10036653-Presyncope (Nervous system disorders) | 1
10044565-Tremor (Nervous system disorders) | 1
10002855-Anxiety (Psychiatric disorders) | 13
10012378-Depression (Psychiatric disorders) | 10
10022437-Insomnia (Psychiatric disorders) | 15
10019450-Hematuria (Renal and urinary disorders) | 2
10037032-Proteinuria (Renal and urinary disorders) | 1
10046539-Urinary frequency (Renal and urinary disorders) | 5
10046543-Urinary incontinence (Renal and urinary disorders) | 3
10046555-Urinary retention (Renal and urinary disorders) | 1
10046593-Urinary urgency (Renal and urinary disorders) | 3
10046628-Urine discoloration (Renal and urinary disorders) | 1
10062225-Urinary tract pain (Renal and urinary disorders) | 1
10006298-Breast pain (Reproductive system and breast disorders) | 4
10022992-Irregular menstruation (Reproductive system and breast disorders) | 1
10036601-Premature menopause (Reproductive system and breast disorders) | 1
10046901-Vaginal discharge (Reproductive system and breast disorders) | 2
10046904-Vaginal dryness (Reproductive system and breast disorders) | 1
10046912-Vaginal hemorrhage (Reproductive system and breast disorders) | 1
10001723-Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5
10011224-Cough (Respiratory, thoracic and mediastinal disorders) | 6
10013963-Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
10015090-Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
10028735-Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
10036402-Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2
10036790-Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
10041232-Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
10041367-Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
10047924-Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
10001760-Alopecia (Skin and subcutaneous tissue disorders) | 40
10013786-Dry skin (Skin and subcutaneous tissue disorders) | 2
10020642-Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
10028691-Nail discoloration (Skin and subcutaneous tissue disorders) | 7
10037087-Pruritus (Skin and subcutaneous tissue disorders) | 2
10037847-Rash acneiform (Skin and subcutaneous tissue disorders) | 10
10037868-Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
10040785-Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 9
10040865-Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 7
10062283-Nail ridging (Skin and subcutaneous tissue disorders) | 2
10027308-Menopause (Social circumstances) | 1
10041244-Social circumstances - Other, specify (Social circumstances) | 1
10016825-Flushing (Vascular disorders) | 1
10019428-Hematoma (Vascular disorders) | 2
10020407-Hot flashes (Vascular disorders) | 14
10020772-Hypertension (Vascular disorders) | 52
10021097-Hypotension (Vascular disorders) | 5
10047065-Vascular disorders - Other, specify (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/66/NCT01525966/Prot_SAP_000.pdf